CLINICAL TRIAL: NCT05213000
Title: The Effect of Health Behavioral Variables Including Single Session Exercise Post-immunization and Psychosocial Factors on Immune Response to the Initial COVID-19 mRNA Vaccine, and Underlying Mechanisms
Brief Title: Adjuvant Effect of Physical Exercise on Immune Response to COVID-19 Vaccination and Interactions With Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Marian Kohut, Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-073
Record Dates: First submitted 2021-10-20; First posted 2022-01-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Immunization
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There are two arms for the initial COVID immunization. The arms are a "control" no exercise group, and an exercise treatment group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise post-immunization (Experimental): After the initial mRNA-based COVID-19 vaccine is received, a supervised 90 minute light to moderate exercise session will take place.
  Interventions: Behavioral: Exercise
- Daily routine as usual (control) (No Intervention): After the initial mRNA-based COVID-19 vaccine is received, participants will be asked to go about their daily routine as usual, but avoid exercise for that day.

INTERVENTIONS:
Behavioral: Exercise — 90 minute exercise session
  Arms: Exercise post-immunization

SUMMARY:
The purpose of this study is to evaluate the extent to which a single session of light to moderate intensity exercise performed within 30 minutes after receiving either the initial dose of COVID-19 mRNA vaccine may modify the immune response to vaccination, and identify potential underlying mechanisms using gene expression and metabolite analysis. A secondary goal is to establish whether psychosocial factors are associated with immune response to vaccination. Participants will be randomized to either a 90-minute light to moderate intensity exercise session or daily routine as usual (no exercise) after receiving their initial COVID-19 mRNA vaccine. If assigned to exercise, the exercise will begin within 30 minutes after receiving the vaccine and will consist of a brisk walk and/or jog supervised by study personnel. Blood will be collected from participants prior the initial dose, two weeks after the initial dose, one week after the second dose if the individual receive the two-dose vaccine regiment or one month after the initial dose if the individual receives a one-dose vaccine regimen, and three, six, and 12 months following the initial dose. . Side effects will be measured for three days post-vaccination. Antibody and cell-mediated immune response to the vaccine will be measured in blood samples. Gene expression profiles will be analyzed by single cell RNA sequencing. Serum metabolites will be assessed to align with immune measures. Participants will be asked to complete surveys to measure physical activity history, psychosocial stress, resilience, and depression. The hypotheses of this study are: 1) a single session of exercise which take place shortly after receiving either the initial dose or the booster dose of COVID-19 will increase antibody and T cell response to the vaccine and will be associated with differentially expressed genes and an altered metabolite profile, and 2) higher levels of reported stress, and lower levels of resilience will be associated with a reduced antibody and T cell response to the vaccine.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the extent to which a single 90-minute session of light to moderate intensity exercise performed within 30 minutes after receiving the initial dose of COVID-19 mRNA vaccine may modify the immune response to vaccination and identify potential underlying mechanisms. A secondary goal is to establish whether psychosocial stress, resilience or depression measures are associated with immune response to vaccination. Participants will be randomly assigned to either an exercise post-vaccine condition (intervention group) or a daily routine as usual but with no exercise condition (control group). Blood samples will be collected from participants before the initial COVID vaccine. At this first visit, participants will be given several psychosocial surveys to complete, the 14-item Perceived Stress Scale , the 25-item Resilience Scale, and the Patient Health Questionnaire. Participants will also be given a copy of local mental health resources. All participants will be asked to complete the psychosocial surveys on the day before or the day of vaccination.

On the day the initial COVID-19 mRNA vaccine is administered, participants assigned to the exercise group will meet with research study personnel within 30 minutes after receiving the vaccine at or near the location at which the vaccine is administered. Participants will begin a light to moderate intensity exercise session consisting of brisk walking, alternating walk/jog, or light jog dependent upon the aerobic fitness level of the participant. The intensity of exercise will be adjusted by heart rate and/or the Borg Rating of Perceived Exertion (RPE) 6-20 scale such that heart rate is approximately 70% of age-adjusted maximal heart rate (220-age), a range between 120-140 beats per minute for most participants, at an RPE of 11 (light) - 13 (somewhat hard). Heart rate and RPE will be monitored approximately every 10 minutes and workload will be adjusted by verbal coaching if necessary. Water and light snacks will be freely available throughout exercise. Participants assigned to the daily routine as usual group will be instructed to continue with their day as typical but to avoid exercise on the day of immunization.

All participants will be given a copy of the appropriate Vaccine Information Fact Sheet and three side effect report forms which list the side effects described in the Vaccine Information sheet. All participants will be asked to record side effects on the appropriate form every 24 hours for the first 72 hours after receiving the initial vaccine. Any concerning side effects are to be reported to study personnel, and the participants will be reminded to report such side effects to their health care provider.

Participants will be asked to return for blood collection seven days, approximately one month, and at three, six, and 12 months following vaccination. Serum from blood samples will be frozen for analysis of serum antibody (anti-receptor binding domain IgG) and neutralizing antibody. Peripheral blood mononuclear cells will be frozen from samples collected at seven days, three or six months post-immunization. The ex vivo functions of Severe Acute Respiratory Syndrome Coronavirus 2 specific T cells specific for dominant epitopes will be evaluated by the assessment of intracellular cytokine production profiles using Severe acute respiratory syndrome coronavirus 2 spike peptide pools. Other peripheral blood mononuclear cells will be reserved for RNA-sequencing (RNA-Seq) analysis. Gene expression will be assessed with RNA-Seq (single cell). The RNA-Seq data analysis will be performed by the Genome Informatics Facility (differential gene expression), GO and Kegg pathway analysis) for comparisons between exercise and control participants. Raman analysis will be used to assess metabolite profile in serum.

The frequency of antigen specific T cells expressing interferon-gamma, tumor necrosis factor alpha, or interleukin-2 or multi-cytokine producing cells, serum antibody and neutralizing antibody will be compared between exercise and control participants. Statistical Package for the Social Sciences (SPSS) software will be used in analyses. As a secondary goal, discovery-based analysis to examine potential effects of psychosocial factors will be performed initially with bivariate analysis of survey scores and immune outcome measures (antibody and T cell cytokines). If a significant correlation between psychosocial survey score and an immune outcome measure is observed, additional follow up with regression model analyses to identify the extent to which separate factors contribute to a given immune outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Able to donate a small amount of blood,
* Planning to receive an initial mRNA Severe Acute Respiratory Distress Syndrome Coronavirus 2 vaccine,
* Between 18-64 years of age,
* Regularly participate in some form of exercise two or more times per week, including at least one session equal to or greater than 50 minutes exercise sessions or walk three or more times per week with at least one session equal to or greater than 50 minutes.
* Can safely perform 90 minutes of light to moderate intensity exercise (walk, walk/jog, or jog) based on American College of Sports Medicine exercise participation guidelines

Exclusion Criteria:

* Currently pregnant
* Weigh less than 110 pounds.
* Presence of any conditions that could significantly impact the ability to exercise safely, or unable to receive the mRNA COVID-19 vaccine
* Taking medication that significantly impact immune response or the presence of an immune disorder.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum antibody | Pre-immunization, and at 2 weeks following the initial immunization, approximately one month, three, six, and twelve months after the initial vaccine
  Change in the total serum anti-receptor binding domain IgG antibody and neutralizing antibody to Severe Acute Respiratory Syndrome Coronavirus 2
Change in T cell response | Time frame with respect to intervention after initial COVID immunization, samples will be assessed approximately one and six months after initial vaccine.
  Antigen-specific T cell immunity
Change in Gene expression profile | Time frame if intervention after initial COVID immunization, approximately one and six months post-immunization.
  Differentially expressed genes between treatment groups
Change in Metabolites | Serum samples collected pre-immunization, if intervention after initial vaccine, two weeks post initial dose, and approximately one month post-immunization.
  Metabolite profiles in serum samples will be assessed

SECONDARY OUTCOMES:
Potential role of psychosocial factors and change in immune response | Serum antibody samples at all time points, and T cell at one week post-immunization
  The potential impact of psychosocial factors (stress, resilience) on antibody and T cell response will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this point, the investigators do not envision sharing individual participant data with other researchers.